CLINICAL TRIAL: NCT03868189
Title: Interest of Ultrasonography in Electroneuromyography: Single-blind Randomised Controlled Clinical Trial
Acronym: US ENMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NIMAO/2018-01/SC-01; 2018-A02872-53 (Other: ANSM)
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2021-08

CONDITIONS: Electromyoneurography
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroneuromyography (Experimental)
  Interventions: Other: Electroneuromyography with ultrasound
- control (Placebo Comparator)
  Interventions: Other: Electroneuromyography without ultrasound

INTERVENTIONS:
Other: Electroneuromyography with ultrasound — Patients whose electroneuromyography examination will be performed using an ultrasound
  Arms: electroneuromyography
Other: Electroneuromyography without ultrasound — Patients whose electroneuromyography examination will be performed without ultrasound (fake tracking)
  Arms: control

SUMMARY:
Echo-nerve tracking during an electroneuromyographic (ENMG) examination by identifying the optimal stimulation site would reduce the stimulation intensities delivered to the patient and thus improve the tolerance of this examination.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring an electroneuromyogram whose indication allows the application of a standard protocol of examination.
* Patient that has given his/her free and informed consent.
* Patient that signed the consent form.
* Patient with an health insurance plan.
* The patient is at least 18 years old (≥).
* he patient is under 80 years old (≤).

Exclusion Criteria:

* Patient with symptoms of neuropathy during the screening.
* Patient whose Neurological severity score (NSS) score is ≥ 3.
* Patient whose neurological examination is abnormal and suggestive of neuropathy.
* Patient presenting a pathology that could cause neuropathy (e.g. diabetes, renal failure, etc.).
* Patient already participating in a category 1 research study (Jardé law).
* Patient in an exclusion period determined by another study.
* Patient under the protection of justice, under guardianship or under curatorship.
* Patient refusing to sign the consent form.
* Patient for which it is impossible to provide information about the study.
* Pregnant patient, parturient, or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Supra-maximal stimulation intensity delivered by stimulation site on sensory nerves | Day 0
  unit : milliampere (mA)

SECONDARY OUTCOMES:
Supra-maximal stimulation intensity delivered by stimulation site on the motor nerves | Day 0
  unit : mA
Sensitivity Amplitude per collection site | Day 0
  unit : microvolts (uV)
Motor Amplitude per collection site | Day 0
  unit : Millivolts (mV)
Total number of explored muscles | Day 0
  unit : number
Number of explored unusual muscles | Day 0
  unit : number
Overall examination time between the beginning of the stimulation and the end of the myography examination | Day 0
  unit : minutes
Average time per explored site (total duration divided by the number of explored nerves and muscles) | Day 0
  unit : minutes
Score of satisfaction | Day 0
  Likert scale that range from 1 ("not satisfied at all ") to 4 ("totally satisfied")
Measurement of felt pain | Day 0
  Analogical visual scale of pain from 1 (no pain) to 100 (maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah COUDRAY, MD, Principal Investigator — Nîmes University Hospital
Locations (2):
- France (2):
  - Nîmes University Hospital, Nîmes
  - CHU Nîmes, Nîmes

REFERENCES:
- [Result] Favier-Archinard C, Leguelinel-Blache G, Dubois F, Le Gall T, Bourquard P, Passemard N, Tora S, Rey A, Rossi M, Chevallier T, Cousin C, Favier M. [Development of a standardized guide for optimizing drug adherence information to be dispensed during a pharmaceutical counseling with a multiple myeloma patient: Initial validation]. Bull Cancer. 2018 May;105(5):475-485. doi: 10.1016/j.bulcan.2017.12.011. Epub 2018 Mar 21. French. PMID 29573809
- [Derived] Laure Inghilleri M, Alonso S, Moron H, Ruiz H, Bastide S, Coudray S. The value of ultrasound-guidance of nerves and muscles for patient tolerance and parameters electrodiagnostic studies. Clin Neurophysiol Pract. 2024 Jan 26;9:78-84. doi: 10.1016/j.cnp.2024.01.003. eCollection 2024. PMID 38357416